CLINICAL TRIAL: NCT03000686
Title: The Effects of GSK2586881 on the Responses to Acute Hypoxia and Exercise
Brief Title: Study of GSK2586881 on Acute Hypoxia and Exercise
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated for technical feasibility, operational considerations and futility in line with pre-specified criteria.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 204987; 2016-002465-55 (EudraCT Number)
Record Dates: First submitted 2016-12-19; First posted 2016-12-22 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
Keywords: GSK2586881, Acute hypoxia, Exercise
MeSH Terms: conditions — Motor Activity | interventions — alunacedase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment sequence AB (Experimental): Subjects will receive GSK2586881 in period 1 and saline placebo in period 2. There will be a washout period of 3-14 days between two treatments
  Interventions: Biological: GSK2586881; Other: Placebo
- Treatment sequence BA (Experimental): Subjects will receive saline placebo in period 1 and GSK2586881 in period 2. There will be a washout period of 3-14 days between two treatments
  Interventions: Biological: GSK2586881; Other: Placebo

INTERVENTIONS:
Biological: GSK2586881 — GSK2586881 will be a clear colorless liquid for IV infusion over 3- 5 mins and will be administered as unit dose 0.8 mg/kg.
Other: Placebo — Normal saline (0.9%) will be administered as a single IV dose infusion over 3 to 5 min.

SUMMARY:
This study is conducted to examine how GSK2586881, a recombinant human ACE2 peptide, modulates the acute hypoxic pulmonary vasoconstriction (HPV) response in healthy volunteers. The study will be single-center, randomized, placebo-controlled and double blind (sponsor open). Subjects will be randomized to receive a single intravenous (IV) dose of GSK2586881 or placebo (saline) in a crossover design. The primary objective of the study is to evaluate the effect of a single IV dose of GSK2586881 on the HPV response in healthy volunteers during exercise under hypoxic conditions. Approximately 35 subjects will be enrolled for a maximum of 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator [in consultation with the Medical Monitor if required] agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Note: Screened subjects with laboratory values outside of the normal range may be repeated once for inclusion into the study at the discretion of the Investigator.
* Screening echocardiogram of good quality, without clinically significant abnormalities, and with mild-moderate tricuspid regurgitation sufficient for the reliable estimation of PASP, as determined by the echocardiography core laboratory or responsible cardiologist. Screening PASP within the normal range according to site standards.
* Subjects have not resided at an altitude >1500 meter (m) for more than 7 days in the last 4 month
* Able to complete all study procedures.
* Any contraindication (orthopedic, cardiac etc.) to perform exercise on a bicycle ergometer.
* Body weight 50 to 100 kilogram (kg) (inclusive).
* Male or female (non Child Bearing Potential): Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until at least five half-lives of study medication OR for a cycle of spermatogenesis following five terminal half-lives after the last dose of study medication. a. Vasectomy with documentation of azoospermia. b. Male condom plus partner use of one of the contraceptive options (Contraceptive subdermal implant, Intrauterine device or intrauterine system, Oral Contraceptive- either combined or progestogen alone, Injectable progestogen, Contraceptive vaginal ring, Percutaneous contraceptive patches). This is an all-inclusive list of those methods that meet the following GSK definition of highly effective: having a failure rate of less than 1% per year when used consistently and correctly and, when applicable, in accordance with the product label. For non-product methods (e.g., male sterility), the investigator determines what is consistent and correct use. The GSK definition is based on the definition provided by the International Conference on Harmonization (ICH).The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test), not lactating, and the following condition applies: Non-reproductive potential defined as, 1. Pre-menopausal females with one of the following (Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy). 2. Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent as described in study protocol which includes compliance with the requirements and restrictions listed in the consent form and in the study protocol.

Exclusion Criteria:

* ALT >1.5x Upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QTc > 450 millisecond (msec.)
* Unable to refrain from prescription or non-prescription drugs, including agents active in the central nervous system, vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication and throughout the study, unless in the opinion of the Investigator and/or GSK Medical Monitor (if needed) the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (approximately 240 milliliter [ml]) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core antibody (HBcAb) should also be excluded.
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 ml within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanover, Lower Saxony, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy participants who met the eligibility criteria entered a 2-period crossover study. Participants were randomized to either placebo or GSK2586881 in each Treatment Period. Total duration of participation was 8 weeks. Study was terminated for technical feasibility, operational considerations and futility in line with pre-specified criteria.
Pre-assignment Details: A total of 48 participants were screened, of which 31 failed screening and 17 (11 participants in Part 1 and 6 in Part 2) were enrolled in the study. The study was conducted at a single center in Germany.
Groups:
- Part 1: Placebo/GSK2586881: Participants were administered a single intravenous (IV) dose of placebo in treatment period 1 followed by a washout of period of up to 14 days. In treatment period 2, participants were administered a single IV dose of 0.8 milligrams per kilogram (mg/kg) GSK2586881. During each period, approximately 30 minutes after administration of study treatment, participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 4000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 70% of maximum oxygen consumption (VO2) uptake on an upright cycle ergometer within the hypoxia chamber for 10 minutes.
- Part 1: GSK2586881/Placebo: Participants were administered a single IV dose of 0.8 mg/kg GSK2586881 in treatment period 1 followed by a washout of period of up to 14 days. In treatment period 2, participants were administered a single IV dose of placebo. During each period, approximately 30 minutes after administration of study treatment, participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 4000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 70% of maximum VO2 uptake on an upright cycle ergometer within the hypoxia chamber for 10 minutes.
- Part 2: Placebo/GSK2586881: Participants were administered a single IV dose of placebo in treatment period 1 followed by a washout of period of up to 14 days. In treatment period 2, participants were administered a single IV dose of 0.8 mg/kg GSK2586881. During each period, approximately 30 minutes after administration of study treatment, participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 5000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 50% of maximum VO2 uptake on a semi-recumbent cycle ergometer within the hypoxia chamber for 10 minutes.
- Part 2: GSK2586881/Placebo: Participants were administered a single IV dose of 0.8 mg/kg GSK2586881 in treatment period 1 followed by a washout of period of up to 14 days. In treatment period 2, participants were administered a single IV dose of placebo. During each period, approximately 30 minutes after administration of study treatment, participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 5000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 50% of maximum VO2 uptake on a semi-recumbent cycle ergometer within the hypoxia chamber for 10 minutes.
Period: Part 1, Period 1 (1 Day)
Arm/Group | Part 1: Placebo/GSK2586881 | Part 1: GSK2586881/Placebo | Part 2: Placebo/GSK2586881 | Part 2: GSK2586881/Placebo
Started | 5 | 6 | 0 | 0
Completed | 5 | 5 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Part 1, Wash-out (Up to 14 Days)
Arm/Group | Part 1: Placebo/GSK2586881 | Part 1: GSK2586881/Placebo | Part 2: Placebo/GSK2586881 | Part 2: GSK2586881/Placebo
Started | 5 | 5 | 0 | 0
Completed | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Period 2 (1 Day)
Arm/Group | Part 1: Placebo/GSK2586881 | Part 1: GSK2586881/Placebo | Part 2: Placebo/GSK2586881 | Part 2: GSK2586881/Placebo
Started | 5 | 5 | 0 | 0
Completed | 5 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Period 1 (1 Day)
Arm/Group | Part 1: Placebo/GSK2586881 | Part 1: GSK2586881/Placebo | Part 2: Placebo/GSK2586881 | Part 2: GSK2586881/Placebo
Started | 0 | 0 | 3 | 3
Completed | 0 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Wash-out (Up to 14 Days)
Arm/Group | Part 1: Placebo/GSK2586881 | Part 1: GSK2586881/Placebo | Part 2: Placebo/GSK2586881 | Part 2: GSK2586881/Placebo
Started | 0 | 0 | 3 | 3
Completed | 0 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Period 2 (1 Day)
Arm/Group | Part 1: Placebo/GSK2586881 | Part 1: GSK2586881/Placebo | Part 2: Placebo/GSK2586881 | Part 2: GSK2586881/Placebo
Started | 0 | 0 | 3 | 3
Completed | 0 | 0 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants-Part 1: All participants who were randomized to either of the two treatment sequences Placebo/GSK2586881 or GSK2586881/Placebo and received a single IV dose of GSK2586881 and placebo in either Treatment period 1 or 2 during Part 1 of the study were included. The treatment periods were separated by a wash-out period of 3 to 14 days.
- All Participants-Part 2: All participants who were randomized to either of the two treatment sequences Placebo/GSK2586881 or GSK2586881/Placebo and received a single IV dose of GSK2586881 and placebo in either Treatment period 1 or 2 during Part 2 of the study were included. The treatment periods were separated by a wash-out period of 3 to 14 days.
- Total: Total of all reporting groups
Arm/Group | All Participants-Part 1 | All Participants-Part 2 | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.2 (4.24) | 29.2 (6.21) | 27.2 (5.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 11 | 6 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - White/Caucasian/European Heritage | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Pulmonary Artery Systolic Pressure (PASP) Measured Via Echocardiography-Part 1
Description: Echocardiograms (Echo) were obtained at indicated time points with the participant resting supine or lying on their left side. PASP was determined by measuring maximal tricuspid regurgitation velocity and applying the modified Bernoulli equation to convert this value into pressure values. Change from Baseline is calculated as the post-dose visit value minus the Baseline value. Analysis was performed using a Bayesian repeated measures model adjusting for: participant-level and period-adjusted Baselines, treatment, time and period. Time by treatment and time by period-adjusted Baseline interactions were included. Participant-level Baseline is the mean of two period-specific Baselines. Period-adjusted Baseline is the difference between the period-specific Baseline and participant-level Baseline for each period. No transformation has been applied to the data. Posterior median and 95% credible interval is presented.
Time Frame: Baseline (Day1, predose) and 15 minutes post-infusion, 60 minutes post-chamber entry, immediately post-exercise and 30 minutes post-chamber exit in each treatment period
Population: Modified Intent-To-Treat Part 1 (mITT1) Population comprised of all participants randomized to Part 1 of the study (planned 4000 meter altitude), excluding those randomized in error. Only those participants with data available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Millimeters of mercury
Groups:
- Part 1: Placebo: Participants were administered a single IV dose of placebo in either treatment period 1 or 2 during Part 1 of the study. During each period, approximately 30 minutes after administration of study treatment, the participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 4000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 70% of maximum VO2 uptake on an upright cycle ergometer within the hypoxia chamber for 10 minutes.
- Part 1: GSK2586881 0.8 mg/kg: Participants were administered a single IV dose of 0.8 mg/kg GSK2586881 in either treatment period 1 or 2 during Part 1 of the study. During each period, approximately 30 minutes after administration of study treatment, the participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 4000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 70% of maximum VO2 uptake on an upright cycle ergometer within the hypoxia chamber for 10 minutes.
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 10
Millimeters of mercury
  15 minutes post-infusion | -0.715 [-3.626 to 2.122] | -0.695 [-3.610 to 2.153]
  60 minutes post-chamber entry | 4.299 [-0.052 to 8.633] | 0.275 [-4.044 to 4.577]
  immediately post-exercise | 1.619 [-5.122 to 8.349] | -0.046 [-6.752 to 6.635]
  30 minutes post-chamber exit | -0.189 [-3.590 to 3.097] | -1.026 [-4.393 to 2.284]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = 0.021, 95% CI 2-sided [-2.249 to 2.295], Standard Deviation 1.1339 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval is presented for 15 minutes post-infusion
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -4.021, 95% CI 2-sided [-9.168 to 1.146], Standard Deviation 2.5923 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval is presented for 60 minutes post-chamber entry
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -1.668, 95% CI 2-sided [-10.576 to 7.231], Standard Deviation 4.4927 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval is presented for immediately post-exercise
Statistical Analysis 4: Comparison: Part 1: Placebo vs Part 1: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -0.824, 95% CI 2-sided [-4.142 to 2.506], Standard Deviation 1.6695 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval is presented for 30 minutes post-chamber exit

2. Primary Outcome: Change From Baseline of PASP Measured Via Echocardiography-Part 2
Description: Echocardiograms were obtained with participant resting supine or lying on their left side. Echo during exercise challenge was conducted with participant on a semi-recumbent cycle ergometer tilted by 30 to 40 degrees. PASP was determined by measuring maximal tricuspid regurgitation velocity and applying modified Bernoulli equation to convert this value into pressure values. Change from Baseline is the post-dose visit value minus Baseline value. Analysis was performed using a Bayesian repeated measures model adjusting for: participant-level and period-adjusted Baselines, treatment, time and period. Time by treatment and time by period-adjusted Baseline interactions were included. Participant-level Baseline is the mean of the two period-specific Baselines. Period-adjusted Baseline is the difference between the period-specific Baseline and participant-level Baseline for each period. No transformation has been applied to the data. Posterior median and 95% credible interval is presented.
Time Frame: Baseline (Day1, predose) and 15 minutes post-infusion, 60 minutes post-chamber entry, 2 minutes post-exercise start and 30 minutes post-chamber exit in each treatment period
Population: mITT Part 2 (mITT2) Population comprised of all participants randomized to Part 2 of the study (planned 5000 meter altitude), excluding those randomized in error. Only those participants with data available at the specified time point were analyzed (represented by n=X, X in category titles).
Measure: Median (95% Confidence Interval); unit: Millimeters of mercury
Groups:
- Part 2: Placebo: Participants were administered a single IV dose of placebo in either treatment period 1 or 2 during Part 2 of the study. During each period, approximately 30 minutes after administration of the study treatment, participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 5000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 50% of maximum VO2 uptake on a semi-recumbent cycle ergometer within the hypoxia chamber for 10 minutes.
- Part 2: GSK2586881 0.8 mg/kg: Participants were administered a single IV dose of 0.8 mg/kg GSK2586881 in either treatment period 1 or 2 during Part 2 of the study. During each period, approximately 30 minutes after administration of the study treatment, participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 5000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 50% of maximum VO2 uptake on a semi-recumbent cycle ergometer within the hypoxia chamber for 10 minutes.
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Millimeters of mercury
  15 minutes post-infusion; n=6, 6 | 2.756 [-0.393 to 5.847] | 2.093 [-1.009 to 5.246]
  60 minutes post-chamber entry; n=6, 6 | 9.399 [4.572 to 14.234] | 6.599 [1.697 to 11.439]
  2 minutes post-exercise start; n=6, 5: number analyzed (Participants) | 6 | 5
  2 minutes post-exercise start; n=6, 5 | 14.665 [8.972 to 20.406] | 14.646 [8.517 to 20.455]
  30 minutes post-chamber exit; n=6, 6 | 4.156 [0.904 to 7.468] | 3.867 [0.592 to 7.174]
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -0.662, 95% CI 2-sided [-5.037 to 3.815], Standard Deviation 2.1933 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Part 2: Placebo vs Part 2: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -2.796, 95% CI 2-sided [-9.729 to 4.027], Standard Deviation 3.4297 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Part 2: Placebo vs Part 2: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -0.018, 95% CI 2-sided [-8.475 to 8.086], Standard Deviation 4.1450 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval is presented for 2 minutes post-exercise start
Statistical Analysis 4: Comparison: Part 2: Placebo vs Part 2: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -0.291, 95% CI 2-sided [-4.960 to 4.386], Standard Deviation 2.3277 — [estimate comment as in outcome 1, analysis 4]

3. Secondary Outcome: Change From Baseline in Renin-angiotensin System (RAS) Peptides-Part 1
Description: Blood samples were collected to analyze RAS peptide biomarkers such as angiotensin II (Ang II), Ang 1-7 and Ang 1-5. Baseline is defined as the measurement taken pre-dose during each treatment period (Day1, pre-dose). Change from Baseline is calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day1, predose) and end of infusion, 15 minutes post-infusion, 15 to 45 minutes post-infusion, 60 minutes post-chamber entry, immediately post-exercise, immediately post-chamber exit and 30 minutes post-chamber exit in each treatment period
Population: mITT1 Population. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Picograms per milliliter
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Picograms per milliliter
  Ang II, End of infusion; n=10, 11 | 0.551 [0.289 to 1.051] | 0.278 [0.149 to 0.522]
  Ang II, 15 minutes post-infusion; n=10, 11 | 0.649 [0.392 to 1.073] | 0.305 [0.155 to 0.602]
  Ang II, 15 to 45 minutes post-infusion; n=10, 11 | 0.661 [0.399 to 1.095] | 0.313 [0.176 to 0.556]
  Ang II, 60 minutes post-chamber entry; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang II, 60 minutes post-chamber entry; n=10, 10 | 0.588 [0.288 to 1.203] | 0.270 [0.140 to 0.521]
  Ang II, immediately post-exercise; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang II, immediately post-exercise; n=10, 10 | 1.379 [0.675 to 2.817] | 0.337 [0.193 to 0.587]
  Ang II, immediately post-chamber exit; n=10,10: number analyzed (Participants) | 10 | 10
  Ang II, immediately post-chamber exit; n=10,10 | 1.001 [0.449 to 2.232] | 0.310 [0.170 to 0.566]
  Ang II, 30 minutes post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang II, 30 minutes post-chamber exit; n=10, 10 | 0.754 [0.366 to 1.553] | 0.263 [0.147 to 0.471]
  Ang 1-7, End of infusion; n=10, 11 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.346 [0.950 to 1.908]
  Ang 1-7, 15 minutes post-infusion; n=10, 11 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.658 [1.179 to 2.331]
  Ang 1-7, 15 to 45 minutes post-infusion; n=10, 11 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.686 [1.032 to 2.755]
  Ang 1-7, 60 minutes post-chamber entry; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang 1-7, 60 minutes post-chamber entry; n=10, 10 | 1.072 [0.916 to 1.254] | 2.615 [1.407 to 4.861]
  Ang 1-7, immediately post-exercise; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang 1-7, immediately post-exercise; n=10, 10 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 3.622 [1.612 to 8.141]
  Ang 1-7, immediately post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang 1-7, immediately post-chamber exit; n=10, 10 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 4.584 [2.015 to 10.431]
  Ang 1-7, 30 minutes post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang 1-7, 30 minutes post-chamber exit; n=10, 10 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.179 [1.285 to 3.695]
  Ang 1-5, End of infusion; n=10, 11 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.489 [0.976 to 2.273]
  Ang 1-5, 15 minutes post-infusion; n=10, 11 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.402 [1.481 to 3.895]
  Ang 1-5, 15 to 45 minutes post-infusion; n=10, 11 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.321 [1.368 to 3.935]
  Ang 1-5, 60 minutes post-chamber entry; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang 1-5, 60 minutes post-chamber entry; n=10, 10 | 1.072 [0.916 to 1.254] | 3.007 [1.269 to 7.123]
  Ang 1-5, immediately post-exercise; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang 1-5, immediately post-exercise; n=10, 10 | 1.094 [0.893 to 1.340] | 5.149 [2.299 to 11.532]
  Ang 1-5, immediately post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang 1-5, immediately post-chamber exit; n=10, 10 | 1.108 [0.879 to 1.396] | 5.991 [2.505 to 14.327]
  Ang 1-5, 30 minutes post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  Ang 1-5, 30 minutes post-chamber exit; n=10, 10 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 3.020 [1.542 to 5.915]

4. Secondary Outcome: Change From Baseline in RAS Peptides-Part 2
Description: Blood samples were collected to analyze RAS peptides such as Ang II, Ang 1-7 and Ang 1-5. Baseline is defined as the measurement taken pre-dose during each treatment period (Day1, pre-dose). Change from Baseline is calculated as post-dose visit value minus Baseline value.
Time Frame: as for outcome 3
Population: mITT2 Population. Only those participants with data available at the specified time points were analyzed (represented by n=X, X in category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Picograms per milliliter
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 4 | 5
Picograms per milliliter
  Ang II, End of infusion; n=4, 5 | 0.603 [0.139 to 2.621] | 0.500 [0.143 to 1.743]
  Ang II, 15 minutes post-infusion; n=4, 5 | 0.564 [0.146 to 2.178] | 0.391 [0.122 to 1.255]
  Ang II, 15 to 45 minutes post-infusion; n=4, 5 | 0.596 [0.140 to 2.536] | 0.391 [0.122 to 1.255]
  Ang II, 60 minutes post-chamber entry; n=4, 5 | 0.532 [0.181 to 1.568] | 0.467 [0.142 to 1.532]
  Ang II, immediately post-exercise; n=4, 5 | 0.447 [0.127 to 1.570] | 0.452 [0.140 to 1.454]
  Ang II, immediately post-chamber exit; n=4, 5 | 0.604 [0.212 to 1.725] | 0.391 [0.122 to 1.255]
  Ang II, 30 minutes post-chamber exit; n=4, 5 | 0.358 [0.060 to 2.151] | 0.472 [0.143 to 1.559]
  Ang 1-7, End of infusion; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.285 [0.640 to 2.581]
  Ang 1-7, 15 minutes post-infusion; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.123 [0.762 to 5.913]
  Ang 1-7, 15 to 45 minutes post-infusion; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.782 [0.659 to 4.821]
  Ang 1-7, 60 minutes post-chamber entry; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.469 [0.844 to 7.229]
  Ang 1-7, immediately post-exercise; n=3, 5: number analyzed (Participants) | 3 | 5
  Ang 1-7, immediately post-exercise; n=3, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.992 [0.833 to 4.763]
  Ang 1-7, immediately post-chamber exit; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.668 [0.644 to 4.319]
  Ang 1-7, 30 minutes post-chamber exit; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.105 [0.865 to 5.123]
  Ang 1-5, End of infusion; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 1.998 [0.814 to 4.901]
  Ang 1-5, 15 minutes post-infusion; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.151 [0.849 to 5.452]
  Ang 1-5, 15 to 45 minutes post-infusion; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.722 [1.222 to 6.063]
  Ang 1-5, 60 minutes post-chamber entry; n=4, 5 | 1.426 [0.461 to 4.417] | 3.053 [0.786 to 11.861]
  Ang 1-5, immediately post-exercise; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.498 [0.814 to 7.673]
  Ang 1-5, immediately post-chamber exit; n=4, 5 | 2.246 [0.481 to 10.493] | 2.417 [0.842 to 6.937]
  Ang 1-5, 30 minutes post-chamber exit; n=4, 5 | 1.000 [NA to NA] — Confidence interval could not be estimated as more than 75% of the values were below lower limit of quantification | 2.561 [1.140 to 5.752]

5. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)-Part 1
Description: SBP and DBP were measured in a semi-supine position after 5 minutes of rest for the participant. Baseline is defined as the measurement taken pre-dose during each treatment period (Day1, pre-dose). Change from Baseline is calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose), 15 to 45 minutes post-infusion, immediately post-exercise and 60 minutes post-chamber exit in each treatment period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Millimeters of mercury
  SBP; 15 to 45 minutes post infusion; n=10, 11 | -1.0 (3.30) | -5.9 (6.88)
  SBP; immediately post-exercise; n=10, 10: number analyzed (Participants) | 10 | 10
  SBP; immediately post-exercise; n=10, 10 | 5.4 (12.89) | -3.0 (14.02)
  SBP; 60 minutes post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  SBP; 60 minutes post-chamber exit; n=10, 10 | -4.0 (4.14) | -6.2 (7.28)
  DBP; 15 to 45 minutes post infusion; n=10, 11 | 0.3 (6.41) | -1.2 (4.24)
  DBP; immediately post-exercise; n=10, 10: number analyzed (Participants) | 10 | 10
  DBP; immediately post-exercise; n=10, 10 | 6.7 (12.40) | 0.3 (7.78)
  DBP; 60 minutes post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  DBP; 60 minutes post-chamber exit; n=10, 10 | 0.0 (7.94) | -1.4 (7.57)

6. Secondary Outcome: Change From Baseline in SBP and DBP-Part 2
Description: as for outcome 5
Time Frame: as for outcome 5
Population: mITT2 Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Millimeters of mercury
  SBP; 15 to 45 minutes post infusion | -3.3 (7.00) | -2.2 (7.36)
  SBP; immediately post-exercise | -9.0 (14.64) | -9.5 (12.85)
  SBP; 60 minutes post-chamber exit | 0.0 (8.94) | -1.5 (4.37)
  DBP; 15 to 45 minutes post infusion | -5.3 (5.39) | -0.8 (8.50)
  DBP; immediately post-exercise | -9.0 (10.75) | -6.0 (8.10)
  DBP; 60 minutes post-chamber exit | 1.5 (9.77) | 3.3 (7.09)

7. Secondary Outcome: Change From Baseline in Heart Rate-Part 1
Description: Heart rate was measured in a semi-supine position after 5 minutes of rest for the participant. Baseline is defined as the measurement taken pre-dose during each treatment period (Day1, pre-dose). Change from Baseline is calculated as the post-dose visit value minus the Baseline value.
Time Frame: as for outcome 5
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Beats per minute
  15 to 45 minutes post infusion; n=10, 11 | -3.6 (4.45) | 1.2 (5.36)
  immediately post-exercise; n=10, 10: number analyzed (Participants) | 10 | 10
  immediately post-exercise; n=10, 10 | 32.0 (7.48) | 37.7 (10.92)
  60 minutes post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  60 minutes post-chamber exit; n=10, 10 | 7.4 (6.33) | 7.7 (7.26)

8. Secondary Outcome: Change From Baseline in Heart Rate-Part 2
Description: as for outcome 7
Time Frame: as for outcome 5
Population: mITT2 Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Beats per minute
  15 to 45 minutes post infusion | -3.7 (3.44) | 0.0 (3.90)
  immediately post-exercise | 11.8 (7.78) | 16.3 (7.37)
  60 minutes post-chamber exit | -1.5 (4.51) | 1.5 (4.42)

9. Secondary Outcome: Change From Baseline in Oxygen Saturation-Part 1
Description: Oxygen saturation was monitored continuously using pulse oximetry. Analysis was performed using a Bayesian repeated measures model adjusting for: participant-level and period-adjusted Baselines, treatment, time and period. Time by treatment and time by period-adjusted baseline interactions were included. Participant-level Baseline is defined as the mean of the two period-specific baselines. Period-adjusted baseline is defined as the difference between the period-specific baseline and participant-level baseline for each period. No transformation has been applied to the data. Non-informative priors used. Baseline is defined as the measurement taken pre-dose during each treatment period (Day1, pre-dose). Change from Baseline is the post-dose visit value minus Baseline value. Posterior median and 95% credible interval is presented.
Time Frame: Baseline (Day 1, pre-dose), 15 minutes post-infusion, 60 minutes post-chamber entry, immediately post-exercise, 30 minutes post-chamber exit in each treatment period
Population: mITT1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (95% Confidence Interval); unit: Percentage of oxygen
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 10
Percentage of oxygen
  15 minutes post-infusion | 1.626 [0.614 to 2.635] | 1.478 [0.467 to 2.493]
  60 minutes post-chamber entry | -10.663 [-13.599 to -7.733] | -11.835 [-14.772 to -8.897]
  immediately post-exercise | -14.257 [-17.397 to -11.109] | -14.426 [-17.590 to -11.279]
  30 minutes post-chamber exit | 0.235 [-0.774 to 1.251] | -0.132 [-1.144 to 0.880]
Statistical Analysis 1: Comparison: Part 1: Placebo vs Part 1: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -0.148, 95% CI 2-sided [-1.264 to 0.973], Standard Deviation 0.5622 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval for oxygen saturation at 15 minutes post-infusion is presented
Statistical Analysis 2: Comparison: Part 1: Placebo vs Part 1: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -1.172, 95% CI 2-sided [-5.271 to 2.942], Standard Deviation 2.0720 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval for oxygen saturation at 60 minutes post-chamber entry is presented
Statistical Analysis 3: Comparison: Part 1: Placebo vs Part 1: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -0.169, 95% CI 2-sided [-4.624 to 4.258], Standard Deviation 2.2351 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval for oxygen saturation immediately post-exercise is presented
Statistical Analysis 4: Comparison: Part 1: Placebo vs Part 1: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -0.367, 95% CI 2-sided [-1.498 to 0.753], Standard Deviation 0.5649 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval for oxygen saturation at 30 minutes post-chamber exit is presented

10. Secondary Outcome: Change From Baseline in Oxygen Saturation-Part 2
Description: as for outcome 9
Time Frame: Baseline (Day 1, pre-dose), 15 minutes post-infusion, 60 minutes post-chamber entry, 2 minutes post-exercise start, 30 minutes post-chamber exit in each treatment period
Population: mITT2 Population
Measure: Median (95% Confidence Interval); unit: Percentage of oxygen
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Percentage of oxygen
  15 minutes post-infusion | 0.644 [-0.602 to 1.892] | 0.847 [-0.416 to 2.090]
  60 minutes post-chamber entry | -23.707 [-26.345 to -21.053] | -19.945 [-22.585 to -17.302]
  2 minutes post-exercise start | -22.399 [-26.372 to -18.415] | -23.433 [-27.400 to -19.484]
  30 minutes post-chamber exit | 1.691 [0.614 to 2.763] | 0.821 [-0.246 to 1.918]
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = 0.203, 95% CI 2-sided [-1.578 to 1.968], Standard Deviation 0.8872 — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Part 2: Placebo vs Part 2: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = 3.760, 95% CI 2-sided [-0.001 to 7.495], Standard Deviation 1.8799 — [estimate comment as in outcome 9, analysis 2]
Statistical Analysis 3: Comparison: Part 2: Placebo vs Part 2: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -1.029, 95% CI 2-sided [-6.673 to 4.578], Standard Deviation 2.8146 — Posterior median difference (GSK2586881 0.8 mg/kg - Placebo) and 95% credible interval for oxygen saturation at 2 minutes post-exercise start is presented
Statistical Analysis 4: Comparison: Part 2: Placebo vs Part 2: GSK2586881 0.8 mg/kg; Test type: Other; Median Difference (Net) = -0.873, 95% CI 2-sided [-2.380 to 0.669], Standard Deviation 0.7620 — [estimate comment as in outcome 9, analysis 4]

11. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings-Part 1
Description: Twelve lead ECGs were obtained using an automated ECG machine that automatically calculated the heart rate and measured PR, QRS, QT and corrected QT (QTc) intervals. ECG was measured in a semi-supine position after 5 minutes rest. Clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings have been presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: pre-dose, 15 to 45 minutes post-infusion, 60 minutes post-chamber exit in each treatment period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Participants
  NCS; pre-dose; n=10, 11 | 8 | 5
  CS; pre-dose; n=10, 11 | 0 | 0
  NCS; 15 to 45 minutes post-infusion; n=10, 11 | 7 | 7
  CS; 15 to 45 minutes post-infusion; n=10, 11 | 0 | 0
  NCS: 60 minutes post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  NCS: 60 minutes post-chamber exit; n=10, 10 | 1 | 3
  CS: 60 minutes post-chamber exit; n=10, 10: number analyzed (Participants) | 10 | 10
  CS: 60 minutes post-chamber exit; n=10, 10 | 0 | 0

12. Secondary Outcome: Number of Participants With Abnormal ECG Findings-Part 2
Description: Twelve lead ECGs were obtained using an automated ECG machine that automatically calculated the heart rate and measured PR, QRS, QT and QTc intervals. ECG was measured in a semi-supine position after 5 minutes rest. Clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings have been presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: pre-dose, 15 to 45 minutes post-infusion, 60 minutes post-chamber exit in each treatment period
Population: mITT2 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Participants
  NCS; pre-dose | 3 | 6
  CS; pre-dose | 0 | 0
  NCS; 15 to 45 minutes post-infusion | 4 | 5
  CS; 15 to 45 minutes post-infusion | 0 | 0
  NCS: 60 minutes post-chamber exit | 3 | 4
  CS: 60 minutes post-chamber exit | 0 | 0

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)-Part 1
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability or incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to 26 days
Population: mITT1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Participants
  AEs | 3 | 2
  SAEs | 0 | 0

14. Secondary Outcome: Number of Participants With AEs and SAEs-Part 2
Description: as for outcome 13
Time Frame: Up to 26 days
Population: mITT2 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Participants
  AEs | 1 | 0
  SAEs | 0 | 0

15. Secondary Outcome: Number of Participants With Positive Immunogenicity Results-Part 1
Description: Blood samples were collected for immunogenicity testing. Blood samples were tested for anti-angiotensin converting enzyme 2 (ACE2) binding antibodies by screening and confirmation assay steps. The post-dose samples tested positive for anti-ACE2 binding antibodies were further characterized for anti-ACE2 neutralizing antibodies. Number of participants with positive incidences for anti-ACE2 binding and neutralizing antibodies is reported.
Time Frame: Up to 26 days
Population: mITT1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

16. Secondary Outcome: Number of Participants With Positive Immunogenicity Results-Part 2
Description: Blood samples were collected for immunogenicity testing. Blood samples were tested for anti-ACE2 binding antibodies by screening and confirmation assay steps. The post-dose samples tested positive for anti-ACE2 binding antibodies were further characterized for anti-ACE2 neutralizing antibodies. Number of participants with positive incidences for anti-ACE2 binding and neutralizing antibodies is reported.
Time Frame: Up to 26 days
Population: mITT2 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

17. Secondary Outcome: Number of Participants With Abnormal Hematology Parameters-Part 1
Description: Blood samples were collected to analyze the following hematology parameters: platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), white blood cell (WBC) count with differential: neutrophils, lymphocytes, monocytes, eosinophils and basophils. Number of participants with abnormal hematology parameters are presented.
Time Frame: Up to 26 days
Population: mITT1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

18. Secondary Outcome: Number of Participants With Abnormal Hematology Parameters-Part 2
Description: Blood samples were collected to analyze the following hematology parameters: platelet count, RBC count, hemoglobin, hematocrit, MCV, MCH, WBC count with differential: neutrophils, lymphocytes, monocytes, eosinophils and basophils. Number of participants with abnormal hematology parameters are presented.
Time Frame: Up to 26 days
Population: mITT2 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

19. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Parameters-Part 1
Description: Blood samples were collected to analyze the following clinical chemistry parameters: blood urea nitrogen (BUN), creatinine, glucose, potassium, sodium, calcium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total and direct bilirubin, total protein and albumin. Number of participants with abnormal clinical chemistry parameters are presented.
Time Frame: Up to 26 days
Population: mITT1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Participants | 0 | 3

20. Secondary Outcome: Number of Participants With Abnormal Clinical Chemistry Parameters-Part 2
Description: Blood samples were collected to analyze the following clinical chemistry parameters: BUN, creatinine, glucose, potassium, sodium, calcium, AST, ALT, alkaline phosphatase, total and direct bilirubin, total protein and albumin. Number of participants with abnormal clinical chemistry parameters are presented.
Time Frame: Up to 26 days
Population: mITT2 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

21. Secondary Outcome: Number of Participants With Abnormal Urine Parameters-Part 1
Description: Urine samples were collected to analyze the following urine parameters: specific gravity, potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick. Microscopic examination was performed for any abnormal dipstick results. Number of participants with abnormal urine parameters are presented.
Time Frame: Up to 26 days
Population: mITT1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

22. Secondary Outcome: Number of Participants With Abnormal Urine Parameters-Part 2
Description: Urine samples were collected to analyze the following urine parameters: specific gravity, pH, glucose, protein, blood and ketones by dipstick. Microscopic examination was performed for any abnormal dipstick results. Number of participants with abnormal urine parameters is presented.
Time Frame: Up to 26 days
Population: mITT2 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

23. Secondary Outcome: Plasma Concentrations of GSK2586881-Part 1
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK2586881. Pharmacokinetic Part1 (PK1) Population comprised of participants in the mITT population, randomized in Part 1 of the study, for whom a pharmacokinetic sample was obtained and analyzed and on active treatment.
Time Frame: pre-dose, at infusion, 15 minutes post-infusion, 15 to 45 minutes post-infusion, 60 minutes post-chamber entry, immediately post-exercise, immediately post-chamber exit and 30 minutes post-chamber exit in each treatment period
Population: PK1 Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles)
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 11
Nanograms per milliliter
  pre-dose; n=11 | NA (NA) — No concentration values detected for pre-dose
  At infusion; n=11 | 10256.935 (2667.2276)
  15 minutes post-infusion; n=11 | 10862.467 (1765.2731)
  15 to 45 minutes post-infusion; n=11 | 9646.325 (1351.1030)
  60 minutes post-chamber entry; n=10: number analyzed (Participants) | 10
  60 minutes post-chamber entry; n=10 | 6934.842 (860.4466)
  immediately post-exercise; n=10: number analyzed (Participants) | 10
  immediately post-exercise; n=10 | 6698.518 (726.7099)
  immediately post-chamber exit; n=10: number analyzed (Participants) | 10
  immediately post-chamber exit; n=10 | 6304.675 (731.1517)
  30 minutes post-chamber exit; n=10: number analyzed (Participants) | 10
  30 minutes post-chamber exit; n=10 | 5209.130 (543.4398)

24. Secondary Outcome: Plasma Concentrations of GSK2586881-Part 2
Description: Blood samples were collected at indicated time points for PK analysis of GSK2586881. Pharmacokinetic Part2 (PK2) Population comprised of participants in the mITT population, randomized in Part 2 of the study, for whom a pharmacokinetic sample was obtained and analyzed and on active treatment.
Time Frame: as for outcome 23
Population: PK2 Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in category titles)
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6
Nanograms per milliliter
  pre-dose; n=5: number analyzed (Participants) | 5
  pre-dose; n=5 | NA (NA) — No concentration values detected for pre-dose
  At infusion; n=6 | 20032.735 (2026.2004)
  15 minutes post-infusion; n=6 | 18269.882 (1790.1483)
  15 to 45 minutes post-infusion; n=6 | 17484.102 (1374.5418)
  60 minutes post-chamber entry; n=6 | 11617.538 (1572.8006)
  immediately post-exercise; n=6 | 11818.457 (1950.1873)
  immediately post-chamber exit; n=6 | 10956.927 (1319.8536)
  30 minutes post-chamber exit; n=6 | 9886.477 (1428.6630)

25. Secondary Outcome: Area Under the Concentration-time Curve Over the Study Period (Pre-dose to 30 Minutes Rest Post Chamber Exit) (AUC[0-2.5 Hours])-Part 1
Description: Blood samples were collected at indicated time points for PK analysis of GSK2586881. The pharmacokinetic parameters were calculated by standard non-compartmental analysis.
Time Frame: as for outcome 23
Population: PK1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10
Hours*micrograms per milliliter | 19.977 (14.3)

26. Secondary Outcome: Area Under the Concentration-time Curve Over the Study Period (Pre-dose to 30 Minutes Rest Post Chamber Exit) (AUC[0-2.5 Hours])-Part 2
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK2 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6
Hours*micrograms per milliliter | 32.400 (9.2)

27. Secondary Outcome: Area Under the Concentration-time Curve Over the Time Period for the Hypoxia Challenge (Immediately Prior to Chamber Entry to Chamber Exit) (AUC [0.5-2 Hours])-Part 1
Description: as for outcome 25
Time Frame: immediately prior to chamber entry, 60 minutes post-chamber entry, immediately post-exercise and immediately post-chamber exit in each treatment period
Population: PK1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 10
Hours*micrograms per milliliter | 12.470 (14.3)

28. Secondary Outcome: Area Under the Concentration-time Curve Over the Time Period for the Hypoxia Challenge (Immediately Prior to Chamber Entry to Chamber Exit) (AUC [0.5-2 Hours])-Part 2
Description: as for outcome 25
Time Frame: as for outcome 27
Population: PK2 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6
Hours*micrograms per milliliter | 18.838 (7.8)

29. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK2586881-Part 1
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK1 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 11
Micrograms per milliliter | 11.296 (17.5)

30. Secondary Outcome: Cmax of GSK2586881-Part 2
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK2 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6
Micrograms per milliliter | 20.343 (6.5)

31. Secondary Outcome: Time to Reach Cmax (Tmax) of GSK2586881-Part 1
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK1 Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 11
Hours | 0.28333 [0.0667 to 0.3833]

32. Secondary Outcome: Tmax of GSK2586881-Part 2
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK2 Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6
Hours | 0.08333 [0.0667 to 0.4667]

33. Secondary Outcome: Apparent Terminal Half-life (T1/2) of GSK2586881-Part 1
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK1 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 11
Hours | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, T1/2 could not be estimated.

34. Secondary Outcome: T1/2 of GSK2586881-Part 2
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK2 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6
Hours | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, T1/2 could not be estimated

35. Secondary Outcome: Clearance for GSK2586881-Part 1
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK1 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour per kilogram
Arm/Group | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 11
Liters per hour per kilogram | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, clearance could not be estimated

36. Secondary Outcome: Clearance for GSK2586881-Part 2
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK2 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour per kilogram
Arm/Group | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6
Liters per hour per kilogram | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, clearance could not be estimated

37. Secondary Outcome: Volume of Distribution for GSK2586881-Part 1
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK1 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per kilogram
Arm/Group | Part 1: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 11
Liters per kilogram | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, volume of distribution could not be estimated

38. Secondary Outcome: Volume of Distribution for GSK2586881-Part 2
Description: as for outcome 25
Time Frame: as for outcome 23
Population: PK2 Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per kilogram
Arm/Group | Part 2: GSK2586881 0.8 mg/kg
Number analyzed (Participants) | 6
Liters per kilogram | NA (NA) — The terminal elimination phase could not be identified from the concentration-time profile over the study period; hence, volume of distribution could not be estimated

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected up to 26 days for Part 1 and Part 2
Description: Non-serious AEs and SAEs were collected in mITT1 Population for Part 1 and mITT2 Population for Part 2.
Groups:
- Part 1: GSK2586881: Participants were administered a single IV dose of 0.8 mg/kg GSK2586881 in either treatment period 1 or 2 during Part 1 of the study. During each period, approximately 30 minutes after administration of study treatment, the participants entered the hypoxia chamber and were inside the chamber for approximately 80 minutes, during which they were under the full 4000 meters ± 10% hypoxic conditions. Participants then performed an exercise challenge at 70% of maximum VO2 uptake on an upright cycle ergometer within the hypoxia chamber for 10 minutes.
Arm/Group | Part 1: Placebo | Part 1: GSK2586881 | Part 2: Placebo | Part 2: GSK2586881 0.8 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/10 | 2/11 | 1/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Placebo (N=10) | Part 1: GSK2586881 (N=11) | Part 2: Placebo (N=6) | Part 2: GSK2586881 0.8 mg/kg (N=6)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03000686/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT03000686/SAP_001.pdf